CLINICAL TRIAL: NCT06933914
Title: An Open Label, Multicenter Study to Evaluate the Long-term Safety and Tolerability of MY008211A Tablets in Patients With PNH Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Long-term Safety and Tolerability of MY008211A Tablets in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY008211A-PNH-2-03
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY008211A tablets (Experimental): MY008211A tablets 400mg BID
  Interventions: Drug: MY008211A tablets

INTERVENTIONS:
Drug: MY008211A tablets — Participants will receive MY008211A at a dose of 400 mg orally b.i.d

SUMMARY:
This is a multicenter, single-arm, open-label study to characterize long-term safety and tolerability of MY008211A tablets and to provide access to MY008211A tablets to patients with PNH who have completed Phase 2 or 3 studies with MY008211A tablets.

DETAILED DESCRIPTION:
The purpose of this open-label, single arm, multicenter study is to evaluate the long-term safety, tolerability and efficacy of MY008211A tablets in patients with PNH and to provide access to patients who have completed (without tapering down) Phase 2 and Phase 3 trials and derived benefit from MY008211A treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have previously received and completed MY008211A study treatment, and are judged by the investigator to have treatment benefit and may benefit from continued treatment of MY008211A.
2. Prior vaccinations against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections.

Exclusion Criteria:

1. History of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus.
2. Known or suspected hereditary complement deficiency.
3. Any comorbidity or medical condition (including but not limited to any active systemic bacterial, viral or fungal infection or malignancy) that, in the opinion of the investigator, could put the subject at increased risk or potentially confound study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with adverse events, safety laboratory parameters, vital signs, ECG. | About 100 weeks
  Safety evaluations including but not limited to adverse events, laboratory parameters, vital signs, ECG through End of Study visit every 12 weeks.

SECONDARY OUTCOMES:
Proportion of participants achieving sustained hemoglobin levels ≥ 120 g/L in the absence of red blood cell transfusions | About 100 weeks
  Proportion of participants achieving sustained hemoglobin levels ≥ 120 g/L in the absence of red blood cell transfusions evaluated every 12 weeks.
Change From Baseline in Hemoglobin | About 100 weeks
  Change in hemoglobin concentration from baseline in patients without RBC transfusion every 12 weeks.
The proportion of patients without RBC transfusion. | About 100 weeks
  The proportion of patients without RBC transfusion.
The Clinical BTH Rate | About 100 weeks
  The Clinical BTH Rate
The Major Adverse Vascular Events Rate | About 100 weeks
  The Major Adverse Vascular Events Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Hematology Hospital (Institute of Hematology, Chinese Academy of Medical Sciences), Tianjin, Tianjin Municipality, China